CLINICAL TRIAL: NCT00030511
Title: A Phase II Study of Chronomodulated Preoperative Infusional Chemoradiation for Biliary Tract Cancer
Brief Title: Radiation Therapy and Fluorouracil Before Surgery in Treating Patients With Primary or Recurrent Bile Duct Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-05991; EORTC-05991
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Extrahepatic Bile Duct Cancer; Liver Cancer
Keywords: localized resectable adult primary liver cancer; recurrent adult primary liver cancer; localized extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Fluorouracil; Radiotherapy

INTERVENTIONS:
Drug: fluorouracil
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of combining radiation therapy with fluorouracil before surgery in treating patients who have primary or recurrent bile duct cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pathologic response rate in patients with primary or recurrent biliary duct carcinoma treated with neoadjuvant radiotherapy and fluorouracil followed by surgical resection.
* Determine the tumor response, morbidity, failure patterns (locoregional vs distant), and survival in patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy once daily five days a week for 5.5 weeks. Patients receive fluorouracil IV over 12 hours each day radiotherapy is administered. Four to six weeks after completion of chemoradiotherapy, patients undergo surgical resection. Patients with residual disease after resection may undergo boost radiotherapy.

Patients are followed every 12 weeks until disease progression and then every 16 weeks after disease progression.

PROJECTED ACCRUAL: A total of 20-47 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary or recurrent biliary duct carcinoma from the proximal, middle, or distal bile ducts
* Measurable or evaluable disease that is considered resectable
* No distant metastases

  * No non-contiguous liver metastases
  * Resectable extension into adjacent liver allowed
  * No metastasis to peritoneal cavity
  * No Bismuth type 4 lesion or metastasis to celiac axis or para-aortic lymph nodes
* No tumor encasement of portal vein or hepatic artery
* No gross ascites

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* No cirrhosis
* No active cholangitis
* No fever or signs of infection in biliary drainage system
* Measurement of C-reactive protein optimal
* Bilirubin less than 3 mg/dL

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective barrier contraception during and for 3 months after study
* No weight loss greater than 20% ideal body weight
* No active duodenal or gastric ulcers
* No other prior or concurrent primary malignancy except adequately treated carcinoma in situ of the cervix or basal cell carcinoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 4 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyvin A. Rich, MD, Study Chair — University of Virginia
Locations (6):
- Cancer Center at the University of Virginia, Charlottesville, Virginia, United States
- Belgium (2):
  - Hopital de Jolimont, Haine-Saint-Paul
  - Les Cliniques Saint-Joseph ASBL, Liège
- France (3):
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Cochin, Paris
  - Hopital Paul Brousse, Villejuif